CLINICAL TRIAL: NCT02922686
Title: Oral Flucloxacillin Alone Versus Flucloxacillin and Phenoxymethylpenicillin for the Emergency Department Outpatient Treatment of Cellulitis: a Non-inferiority Randomised Controlled Trial.
Brief Title: Penicillin for the Emergency Department Outpatient Treatment of CELLulitis
Acronym: PEDOCELL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT Number: 2016-001528-69; HRB HRA Project ID (Other Grant/Funding Number: HRA-DI-2015-1297)
Record Dates: First submitted 2016-08-09; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-07

CONDITIONS: Cellulitis; Wound Infection; Abscess
MeSH Terms: conditions — Cellulitis; Wound Infection; Abscess | interventions — Floxacillin; Penicillin V

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- flucloxacillin + phenoxymethylpenicillin (Active Comparator): Flucloxacillin 500 mg four times daily + Phenoxymethylpenicillin 500 mg four times daily for 7 days.
  Interventions: Drug: Flucloxacillin; Drug: Phenoxymethylpenicillin
- flucloxacillin + placebo (Placebo Comparator): Flucloxacillin 500 mg four times daily + Placebo four times daily for 7 days.
  Interventions: Drug: Flucloxacillin; Drug: Placebo (for phenoxymethylpenicillin)

INTERVENTIONS:
Drug: Flucloxacillin — One flucloxacillin capsule of 500mg strength taken four times daily for 7 days
  Other Names: Floxapen, 500 mg Capsules,; Marketing Authorisation Number PA1380/011/002
Drug: Phenoxymethylpenicillin — One capsule of phenoxymethylpenicillin of 500 mg strength taken four times daily for 7 days
  Other Names: Marketing Authorisation Number PL; 04520/0005
  Arms: flucloxacillin + phenoxymethylpenicillin
Drug: Placebo (for phenoxymethylpenicillin) — Over-encapsulation of phenoxymethylpenicillin will be performed by the manufacturer of the investigational medicinal products such that placebo and active phenoxymethylpenicillin are identical in size, shape, colour and smell, and are packaged in identical bottles
  Other Names: Over-encapsulated investigative medicinal product.
  Arms: flucloxacillin + placebo

SUMMARY:
The main objective of this study is to investigate the non-inferiority of oral flucloxacillin alone compared with a combination of oral flucloxacillin and phenoxymethylpenicillin for the emergency department directed outpatient treatment of cellulitis, wound infections and abscesses, recently renamed by the Food and Drug Administration (FDA) as acute bacterial skin and skin structure infections (ABSSSIs). Half of the trial participants will receive flucloxacillin and placebo in combination, and the remaining half will be treated will flucloxacillin and phenoxymethylpenicillin.

In a secondary objective the trial aims to measure adherence and persistence of trial patients with outpatient antibiotic therapy. In addition a within-trial evaluation of the cost per quality adjusted life year (QALY) gained from the use of oral flucloxacillin compared with combination therapy from the perspective of the health-care payer (direct costs) the patient and government. Finally the study will externally validate the Extremity Soft Tissue Infection-score, a Health Related Quality of Life (HRQL) questionnaire designed to quantify the impact of cellulitis, wound infections and abscesses on patient HRQL in clinical trials.

DETAILED DESCRIPTION:
There is obvious clinical equipoise between the use of oral flucloxacillin alone or combined with phenoxymethylpenicillin for the emergency department treatment of cellulitis, wound infections and abscesses as evidenced by current disparate prescribing practice and hospital guidelines. Feasibility studies for the planned trial have shown that 45-50% of emergency department patients with these infections in Ireland are discharged on oral antibiotics which is consistent with findings in other jurisdictions. Despite the significant healthcare and economic costs associated with cellulitis, there is a paucity of scientific evidence concerning the appropriate antibiotic treatment for these conditions. Additionally, "less severe" infections tend to be over-treated and severe infections under-treated, indicating unjustifiable levels of antibiotic misuse, insufficient knowledge of therapeutics and a lack of evidence to risk-stratify patients with cellulitis to different treatments.The planned trial is therefore likely to be definitive due to the current clinical equipoise between the use of both penicillins for the emergency department outpatient treatment of this group of infections

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed cellulitis, wound infections or abscess (ABSSSI) affecting any body part, excluding the perineum, and having any two of the following signs:

  * Erythema
  * Warmth
  * Tenderness / Pain of affected area
  * Oedema / Induration
  * Regional lymphadenopathy
* Cellulitis, wound infection and abscess deemed treatable with oral outpatient antibiotics in which either combination of antibiotic is likely to produce a clinical response (Eron Class 1-2)
* Written informed consent obtained.
* 16 years of age or older.
* Fluency in written and spoken English.
* Willing to return for study follow-up or to have the research nurse visit their home.
* Willing to receive a telephone call from a study investigator.

Exclusion Criteria:

* Penicillin allergy (self-reported or confirmed).
* Any cellulitis, wound infection and abscess that treating clinicians deem treatable with intravenous (IV) antibiotics.
* Any cellulitis, wound infection and abscess that is more severe than Eron Class 2 (Appendix 2)
* Any cellulitis, wound infection and abscess of the perineal region.
* Patients who have received more than 24 hours of effective antibiotics for the current episode of acute cellulitis, wound infection or abscess
* Any medical condition, based on clinical judgment, that may interfere with interpretation of the primary outcome measures (e.g. chronic skin condition at the lesion site)
* Immunodeficiency from primary or secondary causes (e.g. corticosteroids, chemotherapeutic agents).
* Previous history of renal dysfunction or known chronic kidney disease under care of a nephrologist. - Previous history of liver dysfunction defined as chronically deranged liver function tests elicited from medical notes or history.
* Suspected or confirmed septic arthritis.
* Suspected or confirmed osteomyelitis.
* Infection involving prosthetic material.
* Pregnant or lactating women.
* Patients with a previous history of flucloxacillin- associated jaundice/hepatic dysfunction
* Patients with a previous history of MRSA colonization/infection.
* Patients with lactose intolerance diagnosed by a medical professional

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Investigator-determined clinical response | Test Of Cure visit (Day 14-21 post randomization)
  A trained member of the study team will determine clinical cure at the test of cure visit. This is a clinically-determined response to treatment based on the judgment of the trained member of the study team. Clinical cure will be defined as no treatment failure at any previous visit, and resolution or minimal presence of the erythema, swelling, tenderness, or induration from the baseline assessment, based on the study investigators clinical assessment

SECONDARY OUTCOMES:
Early Clinical Response (ECR) | Day 2-3 post randomization
  Early clinical response is defined as greater than or equal to a 20% reduction in the lesion surface area from that which was measured at enrolment.
Clinical Treatment Failure | Up to 21 days post randomization
  Any patient outcome designated as a clinical treatment failure at any time before and including the test of cure visit, will be categorized as a treatment failure. This commences with the early clinical response visit and includes serial changes in the surface area of the cellulitis lesion (erythema, oedema, tenderness and induration), clinical assessment of progress and health related quality of life measurements.
Adherence to Medication | End of Treatment (EOT) visit Day 8-10 post randomization
  Medication adherence will be measured by counting the number of unused study medication at the end of treatment visit
Adherence to medication using an electronic medication event monitoring system (MEMS®) | Day 2-3 and day 8-10 post randomization and initiation of therapy
  A specific sub-study will be performed measuring adherence and persistence to antibiotic treatment using a MEMS® cap. The cap will be fitted to the dispensed medication bottle. MEMS® caps will be returned with the clinical trials supplies on the follow up visits.medication at the end of treatment visit
Measurement of Health Related Quality of Life | Day 2-3 post-randomization, Day 8-10 post randomization, Day 14 -21 post randomization
  The EuroQol (EQ-5D-5L) will be used to obtain patient reports of health related quality of life and used in the estimation of quality adjusted life years.
Validation of the Extremity Soft Tissue Infections (ESTI)- score | Day 2-3 post-randomization, Day 8-10 post randomization, Day 14 -21 post randomization
  The ESTI will be used to obtain patient reports of health related quality of life and will be mapped on to EQ-5D-5L levels, to assess the accuracy of ESTI for use in cost-effectiveness studies
Cost-effectiveness analysis | Day 14 - 21 post randomization
  Analysis will consist of a within-trial evaluation of the cost QALY for oral flucloxacillin compared with oral flucloxacillin and phenoxymethylpenicillin over a one month time horizon from the perspective of the healthcare payer, the patient and the government. The CE analysis will use resource use data, where costs will be assigned to derive cost and will also use the QALY derived from the EQ5D-5L, to give overall cost per QALY.
Measurement of Health Resource Use | Day 2-3 post-randomization, Day 8-10 post randomization, Day 14 -21 post randomization
  A health economics resource utilization tool is being constructed to collect data on resource use, e.g. direct costs- hospital visits, primary care visits, and indirect costs such as transport and lost work productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Moughty, Principal Investigator — Mater Misericordiae University Hospital; Joseph McKeever, Principal Investigator — Connolly Hospital Blanchardstown; Conor Deasy, Principal Investigator — Department of Emergency Medicine, Cork University Hopsital, Cork; Chris Luke, Principal Investigator — Department of Emergency Medicine, Mercy University, Cork; Abel Wakai, MD FRCEM, Principal Investigator — Department of Emergency Medicine, Beaumont Hospital, Dublin
Locations (5):
- Ireland (5):
  - Department of Emergency Medicine, Connolly Hospital,, Blanchardstown, Dublin
  - Department of Emergency Medicine, Mater Misericordiae University Hospital, Dublin, Dublin
  - Beaumont Hospital,, Dublin, Dublin
  - Department of Emergency Medicine, Mercy University Cork, Cork, Greenville Place
  - Department of Emergency Medicine, Cork University Hospital, Cork, Wilton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quirke M, Saunders J, O'Sullivan R, Milenkovski H, Wakai A. A pilot cross-sectional study of patients presenting with cellulitis to emergency departments. Ir Med J. 2014 Nov-Dec;107(10):316-8. PMID 25556256
- [Background] Dong SL, Kelly KD, Oland RC, Holroyd BR, Rowe BH. ED management of cellulitis: a review of five urban centers. Am J Emerg Med. 2001 Nov;19(7):535-40. doi: 10.1053/ajem.2001.28330. PMID 11698996
- [Background] Kilburn SA, Featherstone P, Higgins B, Brindle R. Interventions for cellulitis and erysipelas. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD004299. doi: 10.1002/14651858.CD004299.pub2. PMID 20556757
- [Background] Storck AJ, Laupland KB, Read RR, Mah MW, Gill JM, Nevett D, Louie TJ. Development of a Health-Related Quality of Life Questionnaire (HRQL) for patients with Extremity Soft Tissue Infections (ESTI). BMC Infect Dis. 2006 Oct 11;6:148. doi: 10.1186/1471-2334-6-148. PMID 17034641
- [Background] Quirke M, O'Sullivan R, McCabe A, Ahmed J, Wakai A. Are two penicillins better than one? A systematic review of oral flucloxacillin and penicillin V versus oral flucloxacillin alone for the emergency department treatment of cellulitis. Eur J Emerg Med. 2014 Jun;21(3):170-4. doi: 10.1097/MEJ.0b013e328360d980. PMID 23542420
- [Derived] Boland F, Quirke M, Gannon B, Plunkett S, Hayden J, McCourt J, O'Sullivan R, Eustace J, Deasy C, Wakai A. The Penicillin for the Emergency Department Outpatient treatment of CELLulitis (PEDOCELL) trial: update to the study protocol and detailed statistical analysis plan (SAP). Trials. 2017 Aug 24;18(1):391. doi: 10.1186/s13063-017-2121-2. PMID 28836993